CLINICAL TRIAL: NCT04005729
Title: Platelet Inhibition With Cangrelor in Comatose Survivors of Out-of-hospital Cardiac Arrest Undergoing Primary Percutaneous Coronary Intervention
Brief Title: Cangrelor in Comatose Survivors of OHCA Undergoing Primary PCI
Acronym: Cangrelor OHCA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Medical Centre Ljubljana (Other)
Collaborators: Chiesi Slovenija, d.o.o. (Industry)
Responsible Party: Principal Investigator, Marko Noc, Clinical Professor, University Medical Centre Ljubljana
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KOIIM-2019-1
Record Dates: First submitted 2019-04-01; First posted 2019-07-02 (Actual); Last update posted 2021-12-03 (Actual); Status verified 2021-12

CONDITIONS: Out-Of-Hospital Cardiac Arrest; Acute Coronary Syndrome
Keywords: cangrelor; P2Y12; out-of-hospital cardiac arrest; induced hypothermia; primary percutaneous coronary intervention
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest; Acute Coronary Syndrome | interventions — cangrelor

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cangrelor + Ticagrelor (Experimental): Bolus of cangrelor (30 mcg/kg) and immediately afterwards a continuous intravenous infusion of 4 mcg/kg/min at the start of the primary percutaneous coronary intervention. Crushed and dissolved ticagrelor tablets (180 mg) will be given via inserted enteral tube.
  Interventions: Drug: Cangrelor 50 MG
- Ticagrelor (No Intervention): Crushed and dissolved ticagrelor tablets (180 mg) will be given via enteral tube (standard care).

INTERVENTIONS:
Drug: Cangrelor 50 MG — 30 mcg/kg bolus, then 4h infusion 4 mcg/kg/min
  Other Names: Kengrexal 50 mg
  Arms: Cangrelor + Ticagrelor

SUMMARY:
The main objective of the trial is to find out if 4-hour continuous infusion of parenteral P2Y12 inhibitor cangrelor at the start of primary percutaneous coronary intervention (PCI) immediately and effectively suppresses platelet activity in comatose survivors of out-of-hospital cardiac arrest (OHCA). Half of the participants will receive the standard care of dual antiplatelet therapy - acetysalicylic acid and ticagrelor tablets via nasogastric or orogastric tube and the other half the standard care with additional cangrelor infusion at the start of the PCI.

DETAILED DESCRIPTION:
Coronary artery disease is an important cause of out-of hospital cardiac arrest (OHCA) and around 80 % of patients after OHCA are comatose. Considering patient's history, details concerning OHCA and ECG changes the decision on urgent cardiac catheterization is made. In case of significant coronary artery stenosis/occlusion on primary percutaneous coronary intervention stent implantation is usually needed. Dual antiplatelet therapy is the cornerstone of stent thrombosis prevention. Patients who are comatose after the return of spontaneous circulation (ROSC) differ from conscious survivors of OHCA because they are not able to take antiplatelet drugs, such as P2Y12 inhibitors, orally. Due to the need for nasogastric/ orogastric tube insertion there is a significant delay until optimal antiplatelet effect is achieved. Furthermore, there are other factors that have an impact on the pharmacokinetics of P2Y12 inhibitors, such as therapeutic hypothermia, gastroparesis, gastrointestinal tract hypoperfusion and platelet hyperreactivity because of systemic inflammatory response syndrome. These characteristics make acute and subacute stent thrombosis more common in comatose OHCA survivors leading to increased morbidity and mortality.

Heparin is the primary anticoagulant drug for comatose patients after OHCA. Antiplatelet therapy consists of intravenous aspirin and P2Y12 inhibitor. Ticagrelor is the most potent of the latter. It is available only as a tablet, which has to be crushed and dissolved and then given via nasogastric or orogastric tube. A recent study by Steblovnik et al. has shown there is an approximately 4-hour gap of inadequate platelet inhibition in comatose OHCA even if the most potent P2Y12 inhibitor ticagrelor is used. Prueller made a retrospective study assessing the addition of intravenous P2Y12 inhibitor cangrelor as a bridge of this gap to standard care. The results showed there is a significant antiplatelet effect when using cangrelor with no added bleeding risk. After literature review no prospective randomised study has been done comparing cangrelor-bridge to standard care with dual antiplatelet therapy (aspirin and ticagrelor).

The investigator's study is a single-blinded, prospective randomised study taking place at University Medical Centre Ljubljana. Thirty comatose survivors of OHCA will be randomised at the start of primary PCI into a test and control group. The control group will receive standard care with intravenous aspirin and dissolved ticagrelor tablets given via enteral tube. The test group patients will receive an additional P2Y12 bridging therapy: a bolus of cangrelor at the start of the PCI (30 mcg/kg) followed by a continuous 4-hour infusion (4 mcg/kg/min). Heparin will be used as per guidelines for a target ACT of 250-300 seconds at the time of PCI. Interventional cardiologist will decide on the use of eptifibatide (GP IIb/IIIa antagonist). Therapeutic hypothermia will be started in the catheterisation laboratory. All patients will be transferred to ICU after the procedure and level of platelet inhibition will be tested 1, 3 and 5 hours after the start of cangrelor infusion with VerifyNow and Multiplate systems. In the control group blood will be drawn at the same time intervals. Further management of patients in both arms will be no different from regular care.

ELIGIBILITY:
Inclusion Criteria:

* age 18 to 70 years
* comatose survivors of out-of-hospital cardiac arrest undergoing primary percutaneous coronary intervention
* treatment with induced therapeutic hypothermia
* no contraindication for dual antiplatelet therapy

Exclusion Criteria:

* pregnancy
* patients without return of spontaneous circulation or patients on ECMO
* history of recent P2Y12 use (last 7 days)
* history of recent vitamin K antagonist or NOAC use (last 14 days)
* active bleeding
* history of transient ischemic attack or cerebral vascular insult
* strong bleeding tendency (Child C liver cirrhosis, stage IV-V chronic renal disease)
* history of allergic reactions to acetylsalicylic acid, heparin or P2Y12 inhibitors
* terminal disease or life expectancy less than 1 year

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2021-11-27 (Actual); Study Completion 2021-11-27 (Actual)

PRIMARY OUTCOMES:
VerifyNow P2Y12Test - Platelet Reactivity | 1 hour after the start of cangrelor infusion/1 hour after the start of PPCI in controls
  Platelet inhibition measured by VerifyNow as P2Y12 reaction units (PRU). Platelet reactivity reflects P2Y12 inhibitor effect with higher PRU values showing low P2Y12 response and lower values decreased platelet reactivity due to the effect of a P2Y12 inhibitor. High on-treatment platelet reactivity was defined as >208 PRU.
VerifyNow P2Y12Test - Platelet Reactivity | 3 hours after the start of cangrelor infusion/3 hours after the start of PPCI in controls
  Platelet inhibition measured by VerifyNow as P2Y12 reaction units (PRU). Platelet reactivity reflects P2Y12 inhibitor effect with higher PRU values showing low P2Y12 response and lower values decreased platelet reactivity due to the effect of a P2Y12 inhibitor. High on-treatment platelet reactivity was defined as >208 PRU.
VerifyNow P2Y12Test - Platelet Reactivity | 5 hours after the start of cangrelor infusion/5 hours after the start of PPCI in controls
  Platelet inhibition measured by VerifyNow as P2Y12 reaction units (PRU). Platelet reactivity reflects P2Y12 inhibitor effect with higher PRU values showing low P2Y12 response and lower values decreased platelet reactivity due to the effect of a P2Y12 inhibitor. High on-treatment platelet reactivity was defined as >208 PRU.
Multiplate ADP test | 1 hour after the start of cangrelor infusion/1 hour after the start of PPCI in controls
  Platelet activation by adenosine diphosphate (ADP) expressed in arbitrary aggregation units (U). P2Y12 inhibitors block ADP receptors and decrease platelet activation by ADP. Higher values mean less effect of P2Y12 inhibitors, lower values mean more effect of P2Y12 inhibitors on platelets. High on-treatment platelet reactivity was defined as >46 U.
Multiplate ADP test | 3 hours after the start of cangrelor infusion/3 hours after the start of PPCI in controls
  Platelet activation by adenosine diphosphate (ADP) expressed in arbitrary aggregation units (U). P2Y12 inhibitors block ADP receptors and decrease platelet activation by ADP. Higher values mean less effect of P2Y12 inhibitors, lower values mean more effect of P2Y12 inhibitors on platelets. High on-treatment platelet reactivity was defined as >46 U.
Multiplate ADP test | 5 hours after the start of cangrelor infusion/5 hours after the start of PPCI in controls
  Platelet activation by adenosine diphosphate (ADP) expressed in arbitrary aggregation units (U). P2Y12 inhibitors block ADP receptors and decrease platelet activation by ADP. Higher values mean less effect of P2Y12 inhibitors, lower values mean more effect of P2Y12 inhibitors on platelets. High on-treatment platelet reactivity was defined as >46 U.
BARC score or the need for discontinuation of cangrelor infusion | During the cangrelor infusion and up to 5 hours after the PCI
  Standardized bleeding definition as described by Bleeding Academic Research Consortium (BARC).
  Type 0: no bleeding.
  1. actionable bleeding, does not require treatment by attending physician.
  2. any overt, actionable sign of hemorrhage plus at least one criteria: (1) requiring nonsurgical, medical intervention, (2) leading to increased level of care, or (3) prompting evaluation.
  3. overt bleeding plus (1) haemoglobin drop of more than 3 g/dL or need for transfusion, (2) cardiac tamponade, (3) requiring surgical intervention, (4) intracranial hemorrhage (does not include microbleeds or hemorrhagic transformation, does include intraspinal), (5) intraocular bleed compromising vision.
  4. CABG-related bleeding (not applicable).
  5. Fatal bleeding: (1) probable - clinically suspicious, (2) definite - overt bleeding or autopsy or imaging confirmation.
  Significant bleeding will be defined as BARC 2, 3 and 5 or the need for discontinuation of cangrelor infusion.

SECONDARY OUTCOMES:
Angiographic result - final TIMI flow | Angiography review within 24 hours of P-PCI (the following day)
  Final angiographic result as evaluated by independent blinded interventional cardiologist. Defined as thrombolysis in myocardial infarction (TIMI) flow at the end of the procedure.
  TIMI 0 flow - absence of any antegrade flow beyond a coronary occlusion TIMI 1 flow - faint antegrade coronary flow beyond the occlusion, with incomplete filling of the distal coronary bed TIMI 2 flow - delayed or sluggish antegrade flow with complete filling of the distal territory TIMI 3 flow - normal flow filling the distal coronary bed completely
  Residual thrombus or peripheral embolization will also be noted.
Rate of stent thrombosis | During index patient hospitalization (at discharge from the hospital, up to 30 days)
  Probable or definitive stent thrombosis according to Academic Research Consortium classification (ARC) of stent thrombosis.
  Definite stent thrombosis - confirmed at angiography or autopsy. Probable stent thrombosis - unexplained death within 30 days after P-PCI or new myocardial infarction in P-PCI vessel territory.
Timing of stent thrombosis | During index patient hospitalization (at discharge from the hospital, up to 30 days)
  Probable or definitive stent thrombosis according to Academic Research Consortium classification (ARC) of stent thrombosis based on timing of events.
  Acute stent thrombosis 0-24 hours after stent implantation Subacute stent thrombosis 24 hours to 30 days after stent implantation
Survival | During index hospitalization (at discharge from the hospital, up to 90 days)
  Survival to discharge from hospital.
Survival (CPC) | During index hospitalization (at discharge from the hospital, up to 90 days)
  Survival to discharge from hospital defined as Cerebral performance category (CPC).
  CPC 1 - good cerebral performance (normal life). Conscious, alert, able to work and lead a normal life.
  CPC 2 - moderate cerebral disability (disabled but independent) CPC 3 - severe cerebral disability (conscious but disabled and dependent) CPC 4 - coma or vegetative state (unconscious) CPC 5 - brain death

CONTACTS AND LOCATIONS:
Overall Officials: Marko Noc, MD PhD, Principal Investigator — University Medical Centre Ljubljana
Locations (1):
- University Medical Centre Ljubljana, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Radsel P, Knafelj R, Kocjancic S, Noc M. Angiographic characteristics of coronary disease and postresuscitation electrocardiograms in patients with aborted cardiac arrest outside a hospital. Am J Cardiol. 2011 Sep 1;108(5):634-8. doi: 10.1016/j.amjcard.2011.04.008. Epub 2011 Jun 14. PMID 21676367
- [Background] Ibanez B, James S, Agewall S, Antunes MJ, Bucciarelli-Ducci C, Bueno H, Caforio ALP, Crea F, Goudevenos JA, Halvorsen S, Hindricks G, Kastrati A, Lenzen MJ, Prescott E, Roffi M, Valgimigli M, Varenhorst C, Vranckx P, Widimsky P; ESC Scientific Document Group. 2017 ESC Guidelines for the management of acute myocardial infarction in patients presenting with ST-segment elevation: The Task Force for the management of acute myocardial infarction in patients presenting with ST-segment elevation of the European Society of Cardiology (ESC). Eur Heart J. 2018 Jan 7;39(2):119-177. doi: 10.1093/eurheartj/ehx393. No abstract available. PMID 28886621
- [Background] Hogberg C, Erlinge D, Braun OO. Mild hypothermia does not attenuate platelet aggregation and may even increase ADP-stimulated platelet aggregation after clopidogrel treatment. Thromb J. 2009 Feb 23;7:2. doi: 10.1186/1477-9560-7-2. PMID 19236702
- [Background] Steblovnik K, Blinc A, Mijovski MB, Fister M, Mikuz U, Noc M. Ticagrelor Versus Clopidogrel in Comatose Survivors of Out-of-Hospital Cardiac Arrest Undergoing Percutaneous Coronary Intervention and Hypothermia: A Randomized Study. Circulation. 2016 Dec 20;134(25):2128-2130. doi: 10.1161/CIRCULATIONAHA.116.024872. No abstract available. PMID 27994027
- [Background] Llitjos JF, Sideris G, Voicu S, Bal Dit Sollier C, Deye N, Megarbane B, Drouet L, Henry P, Dillinger JG. Impaired biological response to aspirin in therapeutic hypothermia comatose patients resuscitated from out-of-hospital cardiac arrest. Resuscitation. 2016 Aug;105:16-21. doi: 10.1016/j.resuscitation.2016.04.027. Epub 2016 May 17. PMID 27224446
- [Background] Pruller F, Bis L, Milke OL, Fruhwald F, Patzold S, Altmanninger-Sock S, Siller-Matula J, von Lewinski F, Ablasser K, Sacherer M, von Lewinski D. Cangrelor Induces More Potent Platelet Inhibition without Increasing Bleeding in Resuscitated Patients. J Clin Med. 2018 Nov 15;7(11):442. doi: 10.3390/jcm7110442. PMID 30445678
- [Background] Mehran R, Rao SV, Bhatt DL, Gibson CM, Caixeta A, Eikelboom J, Kaul S, Wiviott SD, Menon V, Nikolsky E, Serebruany V, Valgimigli M, Vranckx P, Taggart D, Sabik JF, Cutlip DE, Krucoff MW, Ohman EM, Steg PG, White H. Standardized bleeding definitions for cardiovascular clinical trials: a consensus report from the Bleeding Academic Research Consortium. Circulation. 2011 Jun 14;123(23):2736-47. doi: 10.1161/CIRCULATIONAHA.110.009449. No abstract available. PMID 21670242
- [Background] Cutlip DE, Windecker S, Mehran R, Boam A, Cohen DJ, van Es GA, Steg PG, Morel MA, Mauri L, Vranckx P, McFadden E, Lansky A, Hamon M, Krucoff MW, Serruys PW; Academic Research Consortium. Clinical end points in coronary stent trials: a case for standardized definitions. Circulation. 2007 May 1;115(17):2344-51. doi: 10.1161/CIRCULATIONAHA.106.685313. PMID 17470709